CLINICAL TRIAL: NCT00742417
Title: Phase II Study to Evaluate the Efficacy and Safety of Plasma Exchange With 5% Albumin in Beta-amyloid Peptide Clearance in Cerebral Spinal Fluid, and Its Effects in Patients With Mild-moderate Alzheimer's Disease.
Brief Title: Efficacy and Safety of Plasma Exchange With 5% Albumin in Beta-amyloid Peptide Clearance in Cerebral Spinal Fluid
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Instituto Grifols, S.A. (Industry)
Collaborators: Grifols Biologicals, LLC (Industry)
Responsible Party: Sponsor
Organization: Grifols Biologicals, LLC (Industry)
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IG0602
Record Dates: First submitted 2008-08-25; First posted 2008-08-27 (Estimated); Results first posted 2016-06-14 (Estimated); Last update posted 2016-06-14 (Estimated); Status verified 2016-05

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's; Dementia; Senile; Loss of cognitive abilities; Old age; Elderly; Aging; Albumin; Caregiver; amyloid; beta amyloid; Central Nervous System Diseases; Brain Disease; Mental Disorders; Plasma Exchange
MeSH Terms: conditions — Alzheimer Disease; Dementia; Plaque, Amyloid; Central Nervous System Diseases; Brain Diseases; Mental Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Albutein 5% (Experimental): Patients allocated to this arm underwent plasma exchange with Albutein 5%.
  Interventions: Biological: Albutein 5%
- Control (Sham Comparator)
  Interventions: Other: Control

INTERVENTIONS:
Biological: Albutein 5% — 18 Plasma Exchanges using Albutein 5%:
  * three weeks of intensive treatment with two plasma exchanges per week
  * six weeks of maintenance treatment with one weekly plasma exchange
  * three months of maintenance treatment with one plasma exchange every two weeks
  Arms: Albutein 5%
Other: Control — Control group followed the same schedule; however, they did not undergo plasma replacement (it was subjected to simulated plasma replacements)
  Arms: Control

SUMMARY:
The purpose of this study was to evaluate the efficacy and safety of plasma exchange with 5% albumin in beta-amyloid peptide clearance in cerebrospinal fluid, and its effects in patients with mild-moderate Alzheimer's disease.

DETAILED DESCRIPTION:
A phase II study was conducted primarily to determine whether plasma exchange with 5% human albumin is able to modify the concentration of beta-amyloid peptide in cerebrospinal fluid (CSF) in patients with AD.

* There was two weeks for screening and randomization of both groups (treatment and control).
* The subjects were randomized in a 1:1 proportion.

After screening and randomization, treatment proceeded as follows:

* three weeks of intensive treatment with two plasma exchanges per week
* followed by a month and a half of maintenance treatment with one weekly plasma exchange, and
* finally, three months of treatment with one plasma exchange every two weeks.

The control group followed the same program, except for the plasma exchanges. After the treatment period ended, subjects followed-up for a 6-month period of time.

The trial comprises a global multicenter (Spain and US), blind, randomized, controlled design. The trials key coordination is based in Spain where Dr. Boada (see Study Officials/Investigators) is the main study official.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of AD ( National Institute of Neurological and Communicative Disorders and Stroke and the Alzheimer's Disease and Related Disorders Association [NINCDS-ADRDA] criterion), and Mini-mental Status Examination (MMSE) score between ≥18 and ≤26.
* Current stable treatment with acetylcholine esterase inhibitors (AChEIs) for the previous three months.
* A stable care taker must be available, and must attend the patient study visits.
* The patient and a close relative or legal representative must read the patient information sheet, agree to participation in the trial, and then sign the informed consent document (the patient personally and the close relative/legal representative).
* The patient must be able to follow the study protocol, receive the treatment in the established time period, and continue during the follow-up interval.
* A brain Computed Axial Tomography (CAT) or Magnetic Resonance Imaging (MRI) study, obtained in the 12 months prior to recruitment, showing the absence of cerebrovascular disease, must be available.

Exclusion Criteria:

* Any contraindication for plasma exchange due to behavioral disorders or abnormal coagulation parameters
* A history of frequent adverse reactions (serious or otherwise) to blood products.
* Hypersensitivity to albumin or allergies to any of the components of Albutein 5% Human Albumin.
* Plasma creatinine > 2 mg/dL.
* Uncontrolled high blood pressure.
* Liver cirrhosis or any liver problem with alanine aminotransferase (GPT) > 2.5 x upper limit of normal (ULN), or bilirubin > 2 mg/dL.
* Heart diseases, including antecedents of coronary disease and heart failure.
* Difficult venous access precluding plasma exchange.
* Participation in other clinical trials, or the reception of any other investigational drug in the three months prior to the start of the study.
* Any condition complicating adherence to the study protocol (illness with less than one year of expected survival, toxic habits, etc.).
* Pregnant or nursing women or women not using effective contraceptive methods for at least one month after plasma exchange.
* Fewer than six years of education.
* Prior behavioral disorders requiring pharmacological treatment, including insomnia.

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2007-07; Primary Completion 2011-02 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Merce Boada, MD, Principal Investigator — Fundació ACE; Laura Núñez, Study Director — Grifols Biologicals, LLC; Antonio Paez, Study Chair — Grifols Biologicals, LLC
Locations (4):
- United States (2):
  - Howard University, Washington D.C., District of Columbia
  - Mid-Atlantic Geriatric/ARC, Whiting, New Jersey
- Spain (2):
  - Fundació ACE, Barcelona, Catalonia
  - Hospital General Universitario Gregorio Marañon, Madrid, Madrid

RESULTS

PARTICIPANT FLOW:
Groups:
- Control (Sham Procedure): Control group followed the same schedule; however, they did not undergo plasma replacement (it was subjected to simulated plasma replacements)
Period: Randomized
Arm/Group | Albutein 5% | Control (Sham Procedure)
Started | 21 | 21
Completed | 19 | 20
Not Completed | 2 | 1
Not completed — Withdrawal by legal representative | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Physician Decision | 1 | 0
Period: Intensive Period
Arm/Group | Albutein 5% | Control (Sham Procedure)
Started | 19 | 20
Completed | 16 (16 patients completed all the 6 plasma exchange with Albutein 5% during the Intensive Period) | 19 (19 control patients completed all the 6 plasma exchange during the Intensive Period)
Not Completed | 3 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Adverse Event | 2 | 0
Period: Maintenance I
Arm/Group | Albutein 5% | Control (Sham Procedure)
Started | 16 | 19
Completed | 16 | 19
Not Completed | 0 | 0
Period: Maintenance II
Arm/Group | Albutein 5% | Control (Sham Procedure)
Started | 16 | 19
Completed | 16 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The baseline analysis population included all randomized subjects who received at least one plasma exchange session or one sham procedure.
Groups:
- Total: Total of all reporting groups
Arm/Group | Albutein 5% | Control | Total
Number analyzed (Participants) | 19 | 20 | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 10 | 17
  >=65 years | 12 | 10 | 22
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 15 | 30
  Male | 4 | 5 | 9
Weight [Mean (Standard Deviation); unit: Kg] | 64.0 (14.5) | 66.0 (16.6) | 65.1 (15.5)
Height [Mean (Standard Deviation); unit: cm] | 156.8 (11.2) | 159.3 (9.4) | 158.3 (10.1)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Aβ1-42 Cerebrospinal Fluid (CSF) Levels.
Description: Change in levels of Aβ1-42 in CSF in the period between baseline lumbar puncture (before the start of treatment) and lumbar puncture immediately after the end of the last plasma exchange (whenever this may be). Separate assays of Aβ1-42 were performed with Innotest and The Genetics Company commercial kits.
Time Frame: Baseline and up to week 44
Population: The efficacy analyses were performed with the full analysis set (FAS) population which was defined as the set of subjects who were randomized, and received at least three plasma exchange sessions (or sham procedures) during the intensive treatment phase (the three first weeks of treatment).
Measure: Least Squares Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Albutein 5% | Control (Sham Procedure)
Number analyzed (Participants) | 18 | 19
pg/mL
  Aβ1-42 Innotest | 75.3 [-20.0 to 170.5] | -45.5 [-135.1 to 44.2]
  Aβ1-42 The Genetics Company | -86.2 [-253.9 to 81.5] | -283.0 [-441.1 to -125.0]

2. Secondary Outcome: P-Tau and Tau CSF Levels Throughout the Study.
Description: Levels of Tau and P-tau in CSF throughout the treatment phase and the follow-up phase (week 44).
Time Frame: Baseline, week 02, week 08, week 20, week 33 and week 44
Population: The efficacy analyses were performed with the FAS population which was defined as the set of subjects who were randomized and received at least three plasma exchange sessions during the intensive treatment phase (the three first weeks of treatment).
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Albutein 5% | Control (Sham Procedure)
Number analyzed (Participants) | 18 | 19
pg/mL
  P-Tau (baseline) (Albutein n=18; Control n=19) | 87.7 (51.4) | 79.0 (35.1)
  P-Tau (week 02) (n=16; n=19) | 87.5 (43.8) | 94.1 (46.7)
  P-Tau (week 08) (n=15; n=18) | 78.9 (46.3) | 78.0 (41.3)
  P-Tau (week 20) (n=15; n=18) | 88.4 (42.0) | 84.1 (36.8)
  P-Tau (week 33) (n=14; n=15) | 91.9 (57.6) | 78.7 (40.4)
  P-Tau (week 44) (n=14; n=14) | 89.9 (54.5) | 85.1 (46.5)
  Tau (baseline) (n=18; n=19) | 571.2 (354.4) | 589.6 (344.2)
  Tau (week 02) (n=16; n=19) | 669.8 (496.8) | 711.0 (388.8)
  Tau (week 08) (n=15; n=18) | 482.2 (307.4) | 526.3 (326.9)
  Tau (week 20) (n=15; n=18) | 537.1 (253.5) | 555.6 (308.3)
  Tau (week 33) (n=14; n=15) | 539.5 (309.6) | 483.5 (318.5)
  Tau (week 44) (n=14; n=14) | 544.3 (299.4) | 544.1 (347.4)

3. Secondary Outcome: Aβ1-40 Plasma Levels Before and After Each Study Period (The Genetics Company).
Description: Plasma levels of Aβ1-40 before and after the Intensive period, Maintenance period I, Maintenance period II and the Follow-up phase (using The Genetics Company commercial kits).
Time Frame: Baseline, pre-plasma exchange 1 (PRE-PE1), post-plasma exchange 6 (POST-PE6), pre-plasma exchange 7 (PRE-PE7), post-plasma exchange 12 (POST-PE12), pre-plasma exchange 13 (PRE-PE13), post-plasma exchange 18 (POST-PE18), week 33 and week 44.
Population: The efficacy analyses were performed with the FAS population which was defined as the set of subjects who were randomized, and received at least three plasma exchange sessions during the intensive treatment phase (the three first weeks of treatment).
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Albutein 5% | Control
Number analyzed (Participants) | 18 | 19
pg/mL
  Aβ1-40 Baseline (Albutein n=18; Control n=18) | 121.3 (52.6) | 126.7 (43.2)
  Aβ1-40 PRE-PE1 (Intensive) (n=18; n=19) | 120.3 (57.1) | 105.8 (47.7)
  Aβ1-40 POST-PE6 (Intensive) (n=15; n=19) | 255.7 (98.4) | 123.9 (53.7)
  Aβ1-40 PRE-PE7(Maintenance I) (n=14; n=17) | 150.7 (51.3) | 139.7 (41.8)
  Aβ1-40 POST-PE12 (Maintenance I) (n=14; n=18) | 287.1 (98.6) | 150.4 (54.4)
  Aβ1-40 PRE-PE13 (Maintenance II) (n=15; n=19) | 150.0 (66.0) | 129.6 (40.3)
  Aβ1-40 POST-PE18 (Maintenance II) (n=14; n=18) | 245.9 (102.0) | 135.4 (50.2)
  Follow up (33 week) (n=14; n=15) | 153.3 (50.6) | 136.9 (37.3)
  Follow up (44 week) (n=15; n=14) | 146.7 (41.7) | 147.1 (23.4)

4. Secondary Outcome: Aβ1-42 Plasma Levels Before and After Each Study Period (The Genetics Company).
Description: Plasma levels of Aβ1-42 before and after the Intensive period, Maintenance period I, Maintenance period II and the Follow-up phase (using The Genetics Company commercial kits).
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Albutein 5% | Control
Number analyzed (Participants) | 18 | 19
pg/mL
  Aβ1-42 Baseline (Albutein n=18; Control n=18) | 2.8 (9.3) | 33.7 (81.4)
  Aβ1-42 PRE-PE1 (Intensive) (n=18; n=19) | 6.6 (16.3) | 20.9 (58.4)
  Aβ1-42 POST-PE6 (Intensive) (n=15; n=19) | 9.8 (15.6) | 4.9 (11.8)
  Aβ1-42 PRE-PE7 (Maintenance) (n=14; n=17) | 0.0 (0.0) | 4.5 (12.9)
  Aβ1-42 POST-PE12 (Maintenance I) (n=14; n=18) | 10.7 (15.9) | 5.9 (14.3)
  Aβ1-42 PRE-PE13 (Maintenance II) (n=15; n=19) | 6.9 (11.8) | 8.2 (17.2)
  Aβ1-42 POST-PE18 (Maintenance II) (n=14; n=18) | 8.0 (16.7) | 7.1 (14.3)
  Follow up (44 week) (n=15; n=14) | 1.7 (6.6) | 10.2 (18.2)

5. Secondary Outcome: Aβ1-42 Plasma Levels Before and After Each Study Period (Innotest).
Description: Plasma levels of Aβ1-42 before and after the Intensive period, Maintenance period I, Maintenance period II and the Follow-up phase (using Innotest commercial kits).
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Albutein 5% | Control
Number analyzed (Participants) | 18 | 19
pg/mL
  Aβ1-42 Baseline (Albutein n=18; Control n=18) | 40.1 (77.1) | 49.5 (43.7)
  Aβ1-42 PRE-PE1 (Intensive) (n=18; n=19) | 20.4 (21.5) | 33.4 (29.1)
  Aβ1-42 POST-PE6 (Intensive) (n=15; n=19) | 29.1 (23.2) | 45.4 (31.3)
  Aβ1-42 PRE-PE7 (Maintenance I) (n=14; n=17) | 29.5 (30.9) | 58.5 (68.1)
  Aβ1-42 POST-PE12 (Maintenance I) (n=14; n=18) | 25.1 (21.0) | 41.4 (35.5)
  Aβ1-42 PRE-PE13 (Maintenance II) (n=15; n=19) | 36.4 (35.9) | 51.2 (48.3)
  Aβ1-42 POST-PE18 (Maintenance II) (n=14; n=18) | 37.1 (40.9) | 45.3 (42.4)
  Follow up (33 week) (n=14; n=15) | 10.1 (12.9) | 10.2 (16.7)
  Follow up (44 week) (n=15; n=14) | 11.3 (11.4) | 11.7 (20.8)

6. Secondary Outcome: Change From Baseline to Week 44 in Cognitive, Functional and Neuropsychiatric Scores (MMSE, ADAS-Cog, NPS Battery and CSDD)
Description: Change in the cognitive, functional and neuropsychiatric scores and overall development.
  * MMSE: Mini Mental State Examination Score (range = 0 to 30, with lower values indicating impairment)
  * ADAS-Cog: Alzheimer's Disease Assessment Scale, Cognitive Subscale (range = 0 to 70, with higher values indicating impairment)
  * NPS (Neuropsychological battery): •SDMT (Symbol Digit Modalities Test, range = 0 to 110, with lower values indicating impairment), •SVF (Semantic Verbal Fluency Test, with a maximum of 44 words in 60 seconds), •PVF F, A and S (Phonetic Verbal Fluency Test, with a maximum of 44 words in 60 seconds), •BNT (Boston Naming Test, with a maximum of 15 pictures), •RAVLT (Rey Auditory Verbal Learning Test, with 15 words the patient should listen and remind)
  * CSDD (Cornell Scale for Depression in Dementia, 0 = none; 1 =mild or intermittent; 2 = severe)
Time Frame: Change from baseline at week 44
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Albutein 5% | Control (Sham Procedure)
Number analyzed (Participants) | 18 | 19
units on a scale
  MMSE (Albutein n=15; Control n=14) | -1.7 (3.2) | -3.8 (5.9)
  ADAS-Cog (n=15; n=14) | 3.9 (6.2) | 6.6 (10.5)
  NPS (SDMT) (n=15; n=14) | 1.3 (11.2) | -0.5 (2.5)
  NPS (SVF) (n=15; n=14) (n=15; n=14) | 2.5 (3.2) | -0.4 (3.8)
  NPS (PVF(F)) (n=15; n=14) | -0.2 (2.6) | 0.6 (3.8)
  NPS (PVF(A)) (n=15; n=14) | 0.2 (3.4) | 0.2 (3.2)
  NPS (PVF(S)) (n=15; n=14) | 1.1 (1.8) | -0.6 (3.3)
  NPS (BNT) (n=15; n=14) | 1.7 (2.5) | 0.3 (4.1)
  NPS (RAVLT Intermediate 1) (n=15; n=14) | 1.1 (1.9) | -0.1 (2.0)
  NPS (RAVLT Intermediate 2) (n=15; n=14) | 0.3 (1.6) | -1.0 (1.5)
  NPS (RAVLT Intermediate 3) (n=15; n=14) | 0.1 (2.1) | -0.3 (2.0)
  NPS (RAVLT Intermediate 4) (n=15; n=14) | -1.1 (1.8) | -0.9 (2.5)
  NPS (RAVLT Intermediate 5) (n=15; n=14) | -0.3 (2.1) | -1.4 (1.8)
  NPS (RAVLT Delayed) (n=15; n=14) | 0.5 (1.6) | 0.1 (1.0)
  CSDD (patient) (n=10; n=7) | -0.8 (2.9) | -2.1 (5.6)
  CSDD (caregiver) (n=13; n=11) | 1.0 (4.1) | 1.8 (3.7)

7. Secondary Outcome: Change From Baseline to Week 44 in Cognitive, Functional and Neuropsychiatric Scores (ADCS-ADL, NPI, CDR-Sb and ADCS-CGIC).
Description: Change in the cognitive, functional and neuropsychiatric scores and overall development.
  * ADCS-ADL: Alzheimer's Disease Cooperative Study/Activities Of Daily Living (23 questions describing daily activity of the subject and requests the informer to describe the actions or behaviors observed. Increased autonomy associated to higher scores, maximum of 78 points and minimum of 0)
  * NPI: Neuropsychiatric Inventory Questions (12 symptom domains scored by frequency [range=0 to 4, higher values being more frequent] and severity [range=1 to 3, higher values being more severe], total score is sum of frequency x severity of all domains)
  * CDR-Sb: Clinical Dementia Rating (range=0 to 3, higher values being more severe)
  * ADCS-CGIC: Alzheimer's Disease Cooperative Study/Clinical Global Impression of Change (7-point Likert scale, 0=not assessed, 1=marked improvement, 2=moderate improvement, 3=minimal improvement, 4=no change, 5=minimal worsening, 6=moderate worsening and 7=marked worsening)
Time Frame: Change from baseline at week 44
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Albutein 5% | Control (Sham Procedure)
Number analyzed (Participants) | 18 | 19
units on a scale
  ADCS-ADL (Albutein n=15; Control n=14) | -7.1 (11.4) | -4.9 (10.9)
  NPI (total score) (n=15; n=14) | -1.7 (14.1) | -4.0 (13.7)
  NPI (total distress) (n=15; n=14) | -2.1 (7.8) | -3.6 (6.4)
  CDR Sb score (n=15; n=14) | 1.7 (1.5) | 1.4 (3.3)
  ADCS-CGIC (n=15; n=14) | 1.5 (0.7) | 1.2 (1.1)

8. Secondary Outcome: Magnetic Resonance Imaging (MRI) Structural Changes Variations Versus Baseline.
Description: Structural changes in volume of the hippocampus, posterior cingular area, and other associated areas by Magnetic Resonance Imaging (MRI). Three measurements were made (week -2 or -1, 20 and 44). It was measured the variations versus the baseline.
Time Frame: Week 00 (baseline), week 20 and week 44
Population: We analyzed two groups of patients, a treatment group of 20 patients, and a control group, also of 20 patients
Measure: Mean (Standard Deviation); unit: cubic centimetres (cc)
Arm/Group | Albutein 5% | Control (Sham Procedure)
Number analyzed (Participants) | 20 | 20
cubic centimetres (cc)
  Hippocampus L (week 00) | 1.90 (0.41) | 1.91 (0.48)
  Hippocampus L (week 20) | 1.76 (0.45) | 1.85 (0.40)
  Hippocampus L (week 44) | 1.64 (0.43) | 1.76 (0.39)
  Hippocampus R (week 00) | 2.04 (0.41) | 2.14 (0.38)
  Hippocampus R (week 20) | 1.98 (0.41) | 2.07 (0.32)
  Hippocampus R (week 44) | 1.88 (0.35) | 1.96 (0.34)
  Post Cingulate (week 00) | 10.60 (1.34) | 10.38 (0.80)
  Post Cingulate (week 20) | 10.22 (1.58) | 10.39 (0.80)
  Post Cingulate (week 44) | 10.60 (1.48) | 10.23 (1.06)
  Total Intracranial Volume (week 00) | 1034.38 (99.77) | 1064.38 (130.29)
  Total Intracranial Volume (week 20) | 990.31 (83.42) | 1042.70 (119.93)
  Total Intracranial Volume (week 44) | 985.43 (86.10) | 1026.51 (148.43)

9. Secondary Outcome: Variations in Hypoperfusion Based on Single Photon Emission Computed Tomography (SPECT)
Description: Percentage of patients with improved perfusion at the end of the study compared to their initial perfusion. Frontal, parietal and temporal lobes were evaluated from the quantified NeuroGam images. This rendered parametric images showed brain alterations with more than 2 standard deviations with respect to a normal data base. Initial parametric images were compared to the final ones and it was considered perfusion improvement those patients that showed less stretch and/or defect intensity.
Time Frame: End of study
Population: We analyzed two groups of patients, a treatment group of 20 patients, and a control group, also of 20 patients
Measure: Number; unit: percentage of participants
Groups:
- Albutein 5%: Patients allocated to this arm will undergo plasma exchange with Albutein 5%.
  Albutein 5%: 18 Plasma Exchanges using
  * Albutein 5% or
  * Sham Procedure
    * three weeks of intensive treatment with two plasma exchanges per week
    * six weeks of maintenance treatment with one weekly plasma exchange
    * three months of maintenance treatment with one plasma exchange every two weeks
Arm/Group | Albutein 5% | Control
Number analyzed (Participants) | 20 | 20
percentage of participants
  Parietal | 25 | 20
  Temporal | 25 | 10
  Frontal | 5 | 5

ADVERSE EVENTS:
Time Frame: Primary criterion of safety was % of plasma exchange (PE) associated with at least one adverse event (AE) that may be related to the study procedure (adverse reaction).
Description: In addition, global consideration will be made of the percentage PE involving some AE, whether or not related to the procedure. Vital signs, anxiety and restlessness tests and the criterion of the investigator were also used to evaluate patient safety.
Arm/Group | Albutein 5% | Control (Sham Procedure)
Serious Adverse Events (participants affected / at risk) | 3/19 | 2/20
Other Adverse Events (participants affected / at risk) | 18/19 | 14/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Albutein 5% (N=19) | Control (Sham Procedure) (N=20)
Medical device complication (General disorders) | 1 (1) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 0 (0) | 1 (1)
Loss of conscieousness (Nervous system disorders) | 1 (1) | 0 (0)
Partial seizures (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Albutein 5% (N=19) | Control (Sham Procedure) (N=20)
Anemia (Blood and lymphatic system disorders) | 7 (7) | 2 (2)
Ocular hypertension (Eye disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Asthenia (General disorders) | 1 (1) | 0 (0)
Catheter site haemorrage (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 5 (5) | 1 (1)
Nasopharyngitis (Infections and infestations) | 2 (2) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Procedural dizziness (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Muscle haemorrage (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dementia Alzheimer's type (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Aggression (Psychiatric disorders) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 4 (4) | 2 (2)
Confusion state (Psychiatric disorders) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Depressive symptom (Psychiatric disorders) | 1 (1) | 0 (0)
Disinhibition (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Photosensivity reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Bunion operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Urinary cistectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators are free to publish the results after signing the final report. When several papers are published, each one will be mainly prepared by the more experienced investigator who will appear as first author. The rest of co-authors will appear in the order considered opportune by the principal investigator. Sponsor will receive a copy of the manuscript for review at least 30 days prior to submission for publication or presentation of the abstract at some scientific meeting.